CLINICAL TRIAL: NCT03217877
Title: a Multi-center, Open-label, Nationwide Registry-based, Randomized, Pragmatic Trial Comparing 2 Post-PCI Management Strategies in High-risk PCI Patients With Complex Clinical and Lesion Characteristics
Brief Title: Pragmatic Trial Comparing Symptom-Oriented Versus Routine Stress Testing in High-Risk Patients Undergoing Percutaneous Coronary Intervention
Acronym: POST PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AMCCV2017-05
Record Dates: First submitted 2017-07-13; First posted 2017-07-14 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease With Myocardial Infarction
Keywords: noninvasive stress testing; high risk; unstable angina; PCI
MeSH Terms: conditions — Coronary Artery Disease, Autosomal Dominant, 1; Angina, Unstable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Routine stress testing after PCI (Active Comparator)
  Interventions: Diagnostic Test: No Routine stress testing
- Routine stress testing at 9~15 months after PCI (Experimental)
  Interventions: Diagnostic Test: routine stress testing

INTERVENTIONS:
Diagnostic Test: routine stress testing — In the group of routine stress testing group, the preselected functional test (exercise ECG, nuclear stress testing, or stress echocardiography) will be performed at 9~15 months after the procedure according to the practice pattern of each participating center.
  Arms: Routine stress testing at 9~15 months after PCI
Diagnostic Test: No Routine stress testing — In the group of symptom oriented stress testing group, the preselected functional test (exercise ECG, nuclear stress testing, or stress echocardiography) will be performed when chest pain or angina symptom is occured after the procedure according to the practice pattern of each participating center.
  Arms: No Routine stress testing after PCI

SUMMARY:
The primary objective of the POST-PCI trial is to compare the clinical outcomes of a post-percutaneous coronary intervention(PCI) aggressive management strategy of routine noninvasive functional testing to a usual-care strategy of symptom-oriented functional testing in patients with high risk clinical, anatomical, and procedural characteristics who received PCI with contemporary drug-eluting stent and bioresorbable vascular scaffold.

ELIGIBILITY:
Inclusion Criteria:

1. Subject was > 19 years of age.
2. Subjects who underwent successful percutaneous coronary intervention with contemporary drug eluting stent, contemporary Bioresorbable Scaffold or drug eluting balloon at In-stent restenosis (ISR) lesion.
3. Patients must have at least one of the following high-risk clinical, lesion, or procedure-related risk factors.

   3-1. Clinical factors; diabetes, renal insufficiency/failure, enzyme positive acute coronary syndrome (ACS) (STEMI or NSTEMI).

   3-2. Lesion- or procedure-related factors ; left main lesion, bifurcation lesion, ostial lesion, chronic total occlusion lesion, multivessel disease (≥ 2 vessels stented), restenotic lesion, diffuse long lesion (lesion length ≥30 mm or stent length ≥32 mm), or vein bypass graft stented
4. The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

1. Cardiogenic shock at the index admission
2. Subject treated with only bare metal stent or balloon angioplasty during the index procedure.
3. Pregnant and/or lactating women.
4. Concurrent medical condition with a life expectancy of less than 1 years
5. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.

6 Subject was unable to provide written informed consent or participate in long-term follow-up.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
composite of major cardiovascular events | 2 year
  a composite of major cardiovascular events that included death from any cause, myocardial infarction, or hospitalization for unstable angina.

SECONDARY OUTCOMES:
Death | 2 year
Myocardial infarction | 2 year
Unstable angina hospitalization | 2 year
Death or myocardial infarction | 2 year
Any hospitalization | 2 year
  cardiac cause vs. noncardiac cause
Invasive catheterization | 2 year
Repeat revascularization procedure | 2 year
  Repeat revascularization procedure during follow-up; target vs. non-target lesion (or vessel), ischemia-driven vs. not ischemia-driven.

CONTACTS AND LOCATIONS:
Overall Officials: Duk-woo Park, MD, Principal Investigator — Asan Medical Center
Locations (11):
- South Korea (11):
  - Gangwon National Univ. Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Bundang CHA Hospital, Seongnam
  - Seoul National University Bundang hospital, Seongnam
  - Asan Medical Center, Seoul
  - Eulji General Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - The Catholic university of Korea, ST. Vincent's Hospital, Suwon
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Choi Y, Kang DY, Kim H, Lee J, Jo S, Ahn JM, Kim N, Yoon YH, Hur SH, Lee CH, Kim WJ, Kang SH, Park CS, Lee BK, Suh JW, Choi JW, Kim KS, Lee SN, Park SJ, Park DW; POST-PCI Investigators. Role of routine surveillance stress testing in patients with or without imaging-guided or physiology-guided PCI. Heart. 2025 Oct 2:heartjnl-2025-326402. doi: 10.1136/heartjnl-2025-326402. Online ahead of print. PMID 41043864
- [Derived] Lee J, Kang DY, Kim H, Choi Y, Jo S, Ahn JM, Kim S, Yoon YH, Hur SH, Lee CH, Kim WJ, Kang SH, Park CS, Lee BK, Suh JW, Choi JW, Kim KS, Lee SN, Park SJ, Park DW. Routine Stress Testing After PCI in Patients With and Without Acute Coronary Syndrome: A Secondary Analysis of the POST-PCI Randomized Clinical Trial. JAMA Cardiol. 2024 Sep 1;9(9):770-780. doi: 10.1001/jamacardio.2024.1556. PMID 38922632
- [Derived] Lee JM, Kim H, Park YS, Jo HH, Lim SM, Lee J, Choi Y, Kang DY, Ahn JM, Kim S, Yoon YH, Hur SH, Lee CH, Kim WJ, Kang SH, Park CS, Lee BK, Suh JW, Choi JW, Kim KS, Lee SN, Park SJ, Park DW; POST-PCI Investigators. Surveillance Stress Testing After Percutaneous Intervention for Patients With Multivessel or Left Main Coronary Disease. J Am Coll Cardiol. 2024 Mar 5;83(9):890-900. doi: 10.1016/j.jacc.2023.12.027. PMID 38418002
- [Derived] Park DW, Kang DY, Ahn JM, Yun SC, Yoon YH, Hur SH, Lee CH, Kim WJ, Kang SH, Park CS, Lee BK, Suh JW, Yoon JH, Choi JW, Kim KS, Choi SW, Lee SN, Park SJ; POST-PCI Investigators. Routine Functional Testing or Standard Care in High-Risk Patients after PCI. N Engl J Med. 2022 Sep 8;387(10):905-915. doi: 10.1056/NEJMoa2208335. Epub 2022 Aug 28. PMID 36036496